CLINICAL TRIAL: NCT06400745
Title: Contralateral Study of Clareon PanOptix Pro vs. Clareon PanOptix
Brief Title: Clareon PanOptix Pro vs. Clareon PanOptix - Study A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ILQ137-C002-A
Record Dates: First submitted 2024-05-02; First posted 2024-05-06 (Actual); Results first posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Aphakia; Presbyopia
Keywords: Cataract; IOL
MeSH Terms: conditions — Aphakia; Presbyopia; Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Intervention Model Description: Contralateral (split face) study design
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- CPO Pro IOL (Experimental): CPO Pro IOL implanted in the first eye, as randomized. The fellow eye will receive CPO IOL. The second eye surgery will occur approximately 7-14 days after the first eye surgery.
  Interventions: Device: CPO Pro IOL; Device: CPO IOL; Procedure: Cataract surgery
- CPO IOL (Active Comparator): CPO IOL implanted in the first eye, as randomized. The fellow eye will receive CPO Pro IOL. The second eye surgery will occur approximately 7-14 days after the first eye surgery.
  Interventions: Device: CPO Pro IOL; Device: CPO IOL; Procedure: Cataract surgery

INTERVENTIONS:
Device: CPO Pro IOL — Intraocular lens (IOL) implanted in the eye for the visual correction of aphakia in adult patients with less than 1 diopter of preexisting corneal astigmatism in whom a cataractous lens has been removed. The IOL is intended to mitigate the effects of presbyopia on intermediate and near visual acuity while maintaining comparable distance visual acuity.
  Other Names: Clareon PanOptix Pro; Model PXYWT0
Device: CPO IOL — Intraocular lens (IOL) implanted in the eye for the visual correction of aphakia in adult patients with less than 1 diopter of preexisting corneal astigmatism in whom a cataractous lens has been removed. The IOL is intended to mitigate the effects of presbyopia on intermediate and near visual acuity while maintaining distance visual acuity.
  Other Names: Clareon PanOptix; Model CNWTT0
Procedure: Cataract surgery — Extraction of the cataractous lens by phacoemulsification, followed by implantation of the IOL.

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of Clareon™ PanOptix™ Pro Trifocal Intraocular Lens (IOL) compared to Clareon™ PanOptix™ Trifocal IOL.

DETAILED DESCRIPTION:
Subjects will attend 9 scheduled study visits for a total individual duration of participation of approximately 6 months. The primary endpoint will be assessed at the Month 2 follow-up visit. Both eyes of a subject must qualify for enrollment into this study.

ELIGIBILITY:
Key Inclusion Criteria:

* Understand and sign an ethics committee-approved informed consent form;
* Willing and able to attend all scheduled study visits as required by the protocol;
* Planned cataract surgery (both eyes);
* Preoperative corneal astigmatism less that 1.00 diopter in each eye.
* Other protocol-defined inclusion criteria may apply.

Key Exclusion Criteria:

* Women of childbearing potential if currently pregnant, intend to become pregnant during the study, or are breastfeeding;
* Ocular conditions as specified in the protocol;
* Subjects who desire monovision correction.
* Other protocol-defined exclusion criteria may apply.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2024-06-18 (Actual); Primary Completion 2024-12-13 (Actual); Study Completion 2025-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Principal Clinical Trial Lead, Surgical, Study Director — Alcon Research, LLC
Locations (8):
- United States (8):
  - Wolstan & Goldberg Eye Associates, Torrance, California
  - Grosinger, Spigelman & Grey Eye Surgeons, P.C., Bloomfield Hills, Michigan
  - Moyes Eye Center, Kansas City, Missouri
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - Carolina Eyecare Physicians, LLC, Mt. Pleasant, South Carolina
  - Vision for Life, Nashville, Tennessee
  - Houston Eye Associates, Houston, Texas
  - The Eye Institute of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 87 randomized participants, 4 were discontinued after randomization and prior to attempted implantation. This reporting group includes all participants with attempted implantation (83).
Units Other Than Participants: eyes
Groups:
- CPO Pro IOL / CPO IOL: CPO Pro IOL Model PXYWT0 implanted in one eye with CPO IOL Model CNWTT0 implanted in the other eye, as randomized. The second eye surgery occurred approximately 7-14 days after the first eye surgery.
Period: Overall Study
Arm/Group | CPO Pro IOL / CPO IOL
Started | 83; 166 eyes
Implanted With CPO Pro IOL Model PXYWT0 | 83; 166 eyes
Implanted With CPO IOL Model CNWTT0 | 83; 166 eyes
Completed | 83; 166 eyes
Not Completed | 0; 0 eyes

BASELINE CHARACTERISTICS:
Population: All-Implanted Analysis Set
Arm/Group | CPO Pro IOL / CPO IOL
Number analyzed (Participants) | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (7.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 73
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 64
  Black or African American | 12
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 1
  Other | 1
Region of Enrollment [Number; unit: participants]
  United States | 83

OUTCOME MEASURES:

1. Primary Outcome: Mean Monocular Photopic Best Corrected Distance Visual Acuity (BCDVA)
Description: Visual Acuity (VA) was assessed for each eye individually using Early Treatment Diabetic Retinopathy Study (ETDRS) reading charts at a distance of 4 meters from the subject under photopic (well-lit) conditions with correction in place. BCDVA was measured in logarithm Minimum Angle of Resolution (logMAR). LogMAR values typically range from -0.3 (20/10 vision on the Snellen chart) to 1 (20/200 vision), with lower scores indicating better vision.
Time Frame: Month 2 postoperative
Population: All-Implanted Analysis Set
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Groups:
- CPO Pro IOL: CPO Pro IOL Model PXYWT0 implanted in one eye during cataract surgery
- CPO IOL: CPO IOL Model CNWTT0 implanted in one eye during cataract surgery
Arm/Group | CPO Pro IOL | CPO IOL
Number analyzed (Participants) | 83 | 83
Number analyzed (eyes) | 83 | 83
logMAR | 0.032 (0.0919) | 0.023 (0.0813)
Statistical Analysis 1: Comparison: CPO Pro IOL vs CPO IOL; Test type: Non-Inferiority — Study success will be concluded if the upper bound of the one-sided 95.1% confidence interval does not exceed the noninferiority margin of 0.1 logMAR; t-test, 1 sided — The upper boundary of the confidence interval is reported instead of a p-value; The upper bound of the one-sided 95.1% confidence limit will be compared to the margin, 0.10 logMAR; Difference in Means = 0.009, 95.1% CI 1-sided [upper limit 0.0232], Standard Error of Mean 0.0085 — Difference in Means = CPO Pro IOL minus CPO

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from time of consent to study exit, approximately 6 months. AEs were obtained through solicited and spontaneous comments from subjects and through observations by the investigator. "At Risk" population for ocular AEs is reported in units of eyes; all other populations are reported in units of subjects. This analysis population includes all eyes with attempted test or comparator article implantation (successful or aborted after contact with the eye).
Description: All subjects were monitored for serious and other ocular and nonocular AEs. However, the nonocular AE arms were not considered at Risk for ocular adverse event terms as the arms are reporting nonocular-specific AEs. Similarly, the ocular AE arms were not considered at Risk for nonocular adverse event terms as the arms are reporting ocular-specific AEs. All-Cause Mortality was not monitored for the ocular arms.
Groups:
- Pretreatment: Adverse events occurring prior to attempted implantation with the IOL, including ocular adverse events in the second surgical eye that may have occurred prior to second eye attempted implantation.
- CPO Pro IOL Model PXYWT0; CPO IOL Model CNWTT0: Ocular adverse events occurring after attempted implantation with the IOL
- Systemic: Nonocular adverse events occurring after attempted implantation with the IOL (CPO PRO IOL or CPO IOL)
Arm/Group | Pretreatment | CPO Pro IOL Model PXYWT0 | CPO IOL Model CNWTT0 | Systemic
All-Cause Mortality (participants affected / at risk) | 0/83 | 0/0 | 0/0 | 0/83
Serious Adverse Events (participants affected / at risk) | 0/83 | 1/83 | 3/83 | 2/83
Other Adverse Events (participants affected / at risk) | 0/83 | 6/83 | 8/83 | 0/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Pretreatment (N=83) | CPO Pro IOL Model PXYWT0 (N=83) | CPO IOL Model CNWTT0 (N=83) | Systemic (N=83)
Cystoid macular oedema (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0/0
Dry age-related macular degeneration (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0/0
Epiretinal membrane (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0/0
Halo vision (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0/0
Vitreoretinal traction syndrome (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0/0
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0/0 | 0/0 | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0/0 | 0/0 | 1 (1)
Intraocular lens implant (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0/0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Pretreatment (N=83) | CPO Pro IOL Model PXYWT0 (N=83) | CPO IOL Model CNWTT0 (N=83) | Systemic (N=83)
Posterior capsule opacification (Eye disorders) | 0 (0) | 6 (6) | 8 (8) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2025-03-18): https://cdn.clinicaltrials.gov/large-docs/45/NCT06400745/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-04): https://cdn.clinicaltrials.gov/large-docs/45/NCT06400745/SAP_001.pdf